CLINICAL TRIAL: NCT02398955
Title: Biomime Biosorbable Polymer Sirolimus-ELuting Stent in alL-comers patIeNts Treated With Percutaneous Coronary Interventions: the BELLINI Registry
Brief Title: Biomime Stent in All-comers PCI Patients Registry
Acronym: BELLINI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Lupi Alessandro, Dr Alessandro Lupi, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: BELLINI01
Record Dates: First submitted 2015-03-22; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
Keywords: Drug-Eluting Stents; Coronary Artery Disease; Sirolimus; Absorbable Implants
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study cohort: All comers patients with coronary artery disease treated with percutaneous coronary intervention and at least one Biomime stent
  Interventions: Device: percutaneous coronary intervention

INTERVENTIONS:
Device: percutaneous coronary intervention — percutaneous coronary angioplasty with implantation of at least one Biomime stent
  Other Names: Biomime stent

SUMMARY:
Biomime stent is a novel sirolimus-eluting stent (SES) (Meril Life Sciences Pvt. Ltd., Gujarat, India) with an ultra-thin stent platform (65 μm) and a biodegradable polymer licensed for the treatment of de novo coronary lesions. However no data regarding the efficacy and safety of this stent in an "all-comers" patient population treated with percutaneus coronary interventions (PCI) have been published so far. In this registry the investigators aimed to collect clinical and angiographic information about an extensive "all-comers" employ of this novel stent.

ELIGIBILITY:
Inclusion Criteria:

* any coronary artery disease treated with percutaneous coronary intervention and a Biomime stent

Exclusion Criteria:

* patients <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All comers patients with coronary artery disease treated with percutaneous coronary intervention and a Biomime stent, age > 18 years
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
target vessel revascularization | 1 year
  rate of target vessel percutaneous or surgical reintervention for recurrent symptoms or inducible ischemia at follow up testes

SECONDARY OUTCOMES:
death from any cause | 1 year
  death from any cause after the procedure
cardiac death | 1 year
  death form cardiac causes (reinfarction, sudden cardiac death, death during coronary reintervention, heart failure, arrhythmias)
reinfarction | 1 year
  reinfarction in the myocardial region supplied by the treated coronary artery
target lesion revascularization | 1 year
  rate of target lesion percutaneous reintervention for recurrent symptoms or inducible ischemia at follow up testes

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Lupi, MD, Principal Investigator — Azienda Ospedaliero Universitaria Maggiore della Carita
Locations (1):
- Azienda Ospedaliero Universitaria Maggiore della Carita, Novara, Piedmont, Italy